CLINICAL TRIAL: NCT04049422
Title: Pulmonary Nodule Cohort
Acronym: liquidNodule
Status: Not yet recruiting | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Young Sik Park, Associate Professor, Seoul National University Hospital
Other Study IDs: 1907-099-1048
Record Dates: First submitted 2019-08-05; First posted 2019-08-08 (Actual); Last update posted 2019-08-08 (Actual); Status verified 2019-08

CONDITIONS: Pulmonary Nodule, Solitary; Lung Cancer
MeSH Terms: conditions — Solitary Pulmonary Nodule; Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — bronchoalveolar lavage fluid, buffy coat, serum, plasma, urine
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to identify the clinical features of pulmonary nodules and establish a cohort to identify biomarkers for lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* age >= 18
* pulmonary nodule(s) on chest CT, which satisfy at least one of the following two criteria,

  * 4A or above in Lung-RADS v1.1
  * lung cancer risk >= 5% in Brock model

Exclusion Criteria:

* already proven lung cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People with pulmonary nodule(s) for which lung cancer is suspected
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-08-06 (Estimated); Primary Completion 2024-07-31 (Estimated); Study Completion 2029-07-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of lung cancer | up to 5 years
  incidence of pathologically proven lung cancer

IPD SHARING:
Plan to Share IPD: No